CLINICAL TRIAL: NCT07266623
Title: Effects of Muscle Energy Techniques With and Without Manual Axial Distraction on Pain, Range of Motion Anf Functional Outcomes in Post-Mastectomy Patients With Axillary Web Syndrome
Brief Title: Effects of Muscle Energy Techniques With and Without Manual Axial Distraction in Post-Mastectomy Patients With Axillary Web Syndrome
Acronym: MET MAD PM AWS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/031
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Axillary Web Syndrome; Post-mastectomy
Keywords: Axillary web syndrome; Muscle energy techniques; Manual axial distraction; Functional outcomes; Range of motion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, the blinding of participants and therapists was not feasible. To overcome the assessment bias, the outcome assessor remained blinded to group allocations, maintaining single blinded study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Muscle energy technique + Manual axial distraction) (Experimental)
  Interventions: Other: Muscle energy technique + Manual axial distraction
- Group B (Muscle energy technique only) (Experimental)
  Interventions: Other: Muscle energy technique

INTERVENTIONS:
Other: Muscle energy technique + Manual axial distraction — In the MET+ MAD group, a combination of muscle energy techniques and manual axial distraction will be applied on the affected side. The use of MET will target the pectoralis major, supraspinatus, subscapularis, and latissimus dorsi muscles. The participant will contract the targeted muscle for 10 seconds and then relax it. After that, the therapist will stretch that muscle for 10 to 30 seconds, along with manual axial distraction applied to the affected shoulder. The technique of manual axial distraction will employ firm digital pressure combined with distraction at various points over the fibrous band. The intervention will be given 3 times a week for 6 weeks, intensity will be according to the participants' tolerance. Each session will continue for 30 to 40 minutes
  Arms: Group A (Muscle energy technique + Manual axial distraction)
Other: Muscle energy technique — Group B will receive only the muscle energy techniques targeting the pectoralis major, supraspinatus, subscapularis, and lattisimus dorsi muscles on the affected side. The participants will contract the target muscle for 10 seconds and then relax it. After that, the therapist will stretch that muscle for 10 to 30 seconds. The intervention will be given three times a week for six weeks, and each session will continue for 30 to 40 minutes.
  Arms: Group B (Muscle energy technique only)

SUMMARY:
This randomized controlled trial aims to evaluate the effects of muscle energy techniques with and without manual axial distraction among post-mastectomy patients with axillary web syndrome. Fifty-eight participants will be randomly allocated into two groups and will receive the interventions for six weeks. It is hypothesized that the group that will receive both the muscle energy technique and manual axial distraction will produce greater improvements compared to the other group that will receive only MET.

DETAILED DESCRIPTION:
Axillary web syndrome (AWS) is a common post-mastectomy complication characterized by painful, palpable cords that limit shoulder mobility and functional performance. Current rehabilitation approaches emphasize soft-tissue mobilization, stretching, and manual therapy, yet evidence regarding the combined application of muscle energy technique (MET) and manual axial distraction (MAD) remains limited. This randomized controlled trial is designed to compare the effectiveness of MET alone versus MET combined with MAD in improving pain, range of motion (ROM), cord resolution, and functional outcomes in women with AWS. Participants will be randomly assigned to one of two groups using a concealed allocation procedure. All participants will begin each session with a 10-minute heating pad application to promote tissue elasticity, followed by a standardized stretching protocol targeting shoulder flexion and abduction in both supine and sitting positions; each stretch will be repeated five times and held for 30 seconds. The intervention group will receive MET applied to the pectoralis major, supraspinatus, subscapularis, and latissimus dorsi muscles in addition to MAD. MET will be administered using approximately 20% isometric contraction effort without pain, held for 7-10 seconds, followed by therapist-assisted stretching to the new tissue barrier; this cycle will be repeated three times per muscle. Positioning will be adapted for each muscle based on anatomical considerations, such as supine positioning with arm abduction for pectoralis major and subscapularis, or seated positioning for supraspinatus. The MAD technique will be performed using sustained shoulder joint traction for 15-30 seconds combined with firm digital pressure along the fibrous cords until a palpable "snapping" sensation indicates cord release. The comparison group will receive the same stretching and MET protocol without MAD. All interventions will be delivered three times per week for six consecutive weeks, with each session lasting approximately 30-40 minutes and tailored to participant tolerance. Primary outcomes include pain (Numeric Rating Scale), shoulder ROM (goniometry). Secondary outcomes include functional outcome( DASH questionnaire) and cord visibility. Outcome assessments will be conducted at baseline and at six weeks by a blinded assessor. Statistical analysis will include normality testing followed by parametric (paired and independent t-tests, ANOVA) or non-parametric equivalents (Wilcoxon or Mann-Whitney U tests) as appropriate. Effect sizes will be calculated, and significance will be set at p < 0.05. The trial is designed to determine whether adding MAD to MET results in superior improvements in tissue extensibility, pain reduction, ROM enhancement, and functional recovery compared with MET alone, thereby providing evidence-based guidance for rehabilitation of post-mastectomy AWS.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AWS following breast cancer surgery
* Females aged 30 to 60 years old
* Participants must be within 1 month to 2 years post-surgery
* Participants having limited shoulder ROM
* Participants must have completed their post-surgery radiation therapy and chemotherapy minimum of 2-3 weeks

Exclusion Criteria:

* Any previous history of shoulder pathology
* Patients with a cervical problem that radiates pain down the shoulder
* Pregnant females
* Bilateral mastectomy
* Ongoing cancer stage
* Participants with ongoing chemotherapy
* Frozen shoulder

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females
Enrollment: 58 (Estimated)
Dates: Start 2025-12-13 (Estimated); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline: Before intervention 6 weeks post-intervention
  Participants will be asked to rate the pain by using an outcome measure tool, NPRS, a numeric pain rating scale that ranges from 0 to 10. O means no pain, 1-3 means mild pain, 4-6 means moderate pain, 7-10 means severe pain.
Shoulder Range of Motion | Baseline: Before intervention 6 weeks post-intervention
  Shoulder range of motion of the affected side will be measured by using an outcome measure tool, goniometry. Shoulder flexion and abduction ranges will be assessed in the sitting position. Each movement will be performed thrice, and the average values will be analyzed accordingly.

SECONDARY OUTCOMES:
Functional Outcomes | Baseline: Before intervention 6 weeks post-intervention
  Functional outcomes of the participants will be measured by using an outcome measure tool, the DASH (Disabilities of the Arm, Shoulder, and Hand) questionnaire. This questionnaire will assess functional measures that have been asked with 30 different questions regarding the disabilities of the arm, shoulder, and hand, and answers will be recorded as no difficulty to mild, moderate, and severe. Each question has a lowest score of 1, which means there is no difficulty in performing a certain task, and a highest score of 5, indicating that the person is unable to perform the task in question. At least 2 questions must be answered to complete the assessment. Scoring is reported between 0 and 100, with higher disability if scores are high.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Tariq Shafi, Study Chair — Lahore University of Biological and Applied Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koehler LA, Blaes AH, Haddad TC, Hunter DW, Hirsch AT, Ludewig PM. Movement, Function, Pain, and Postoperative Edema in Axillary Web Syndrome. Phys Ther. 2015 Oct;95(10):1345-53. doi: 10.2522/ptj.20140377. Epub 2015 May 14. PMID 25977305
- [Background] Meer TA, Noor R, Bashir MS, Ikram M. Comparative effects of lymphatic drainage and soft tissue mobilization on pain threshold, shoulder mobility and quality of life in patients with axillary web syndrome after mastectomy. BMC Womens Health. 2023 Nov 10;23(1):588. doi: 10.1186/s12905-023-02762-w. PMID 37950230
- [Background] Gonzalez-Rubino JB, Vinolo-Gil MJ, Martin-Valero R. Effectiveness of physical therapy in axillary web syndrome after breast cancer: a systematic review and meta-analysis. Support Care Cancer. 2023 Apr 12;31(5):257. doi: 10.1007/s00520-023-07666-x. PMID 37043039
- [Background] Gonzalez-Rubino JB, Martin-Valero R, Vinolo-Gil MJ. Physiotherapy protocol to reduce the evolution time of axillary web syndrome in women post-breast cancer surgery: a randomized clinical trial. Support Care Cancer. 2025 Mar 28;33(4):326. doi: 10.1007/s00520-025-09373-1. PMID 40153020
- [Background] Sandrin F, Nevola Teixeira LF, Garavaglia M, Gandini S, Simoncini MC, Luini A. The efficacy in shoulder range of motion of a snapping manual maneuver added to a standardized exercise protocol in axillary web syndrome: a randomized controlled trial. Acta Oncol. 2023 Aug;62(8):969-976. doi: 10.1080/0284186X.2023.2241995. Epub 2023 Sep 26. PMID 37750301